CLINICAL TRIAL: NCT03776552
Title: Comparative Effectiveness of a Gradual Weight Loss Program and a Rapid Weight Loss Program (Including a Low Energy Diet) on 1-year Weight Loss in Subjects With Obesity - A Randomized, Parallel-group, Superiority Trial. (The GoLow Study).
Brief Title: Effectiveness of Gradual Versus Rapid Weight Loss
Acronym: GoLow
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital of Vestfold (Other)
Collaborators: Roede AS (Unknown)
Responsible Party: Principal Investigator, Jøran Hjelmesæth, Professor, Head, The Hospital of Vestfold
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GoLow
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor was masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid weight loss (RWL) program (Active Comparator): 16-week rapid weight loss (RWL) program [8-week LED (<1000 kcal/day) - followed by an 8-week gradual increase in energy intake (4 weeks <1300 kcal/day and 4 weeks <1500 kcal/day)] followed by a 36-weight loss maintenance program.
  Interventions: Other: Rapid weight loss (RWL) program
- Gradual weight loss (GWL) program (Active Comparator): 16-week GWL-program (estimated total energy expenditure minus 800-1000 kcal/day) followed by a 36-weight loss maintenance program.
  Interventions: Other: Gradual weight loss (GWL) program

INTERVENTIONS:
Other: Rapid weight loss (RWL) program — 16-week rapid weight loss (RWL) program (8-week low energy diet (LED) followed by 8-week gradual increased energy intake) and a subsequent 36-week weight-maintenance follow-up
  Arms: Rapid weight loss (RWL) program
Other: Gradual weight loss (GWL) program — 16-week gradual weight loss (GWL) program (moderate calorie restriction) and a subsequent 36-week weight-maintenance follow-up
  Arms: Gradual weight loss (GWL) program

SUMMARY:
This randomized controlled trial aims to compare the 1-year effectiveness of an initial rapid weight loss (RWL) program and a gradual weight loss (GWL) program.

DETAILED DESCRIPTION:
A total of at least 286 participants will be randomized to either a 16-week rapid weight loss (RWL) program; [an 8-week low-energy-diet (<1000 kcal/day) - followed by an 8-week gradual increase in energy intake (4 weeks <1300 kcal/day and 4 weeks <1500 kcal/day)], or a 16-week gradual weight loss (GWL) program (controls); [estimated total energy expenditure minus 800-1000 kcal/day]. Thereafter, all participants (both groups) will undergo a 36-week comprehensive weight maintenance program.

ELIGIBILITY:
Inclusion Criteria:

* • Willing and able to give informed consent for participation in the study

  * Living in the eastern part of Norway, mainly Oslo, Buskerud, Vestfold and Akershus
  * Understanding Norwegian language written and spoken easily
  * BMI ≥30.0 kg/m2
  * Stable body weight (<5 kg self-reported weight change) during the last 3 months before inclusion

Exclusion Criteria:

* • Pregnancy and breast-feeding mothers

  * Suspected non-compliance with regards to visits and/or diet
  * Severe chronic disease (endocrine disease, heart disease, neurological disease, lung disease, disease in the gastrointestinal tract, kidney disease, rheumatism or cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight from baseline to 12 months | Baseline to 1-year
  Percent total body weight loss (%TBWL) at 12 months follow-up

SECONDARY OUTCOMES:
Changes in anthropometric measures | 4-month and 1-year
  Waist and hip circumference (cm)
Changes in body composition 1 | 4-month and 1-year
  Bioelectrical Impedance Analysis (BIA)
Changes in body composition 2 | 4-month and 1-year
  Dual-energy X-ray Absorptiometry (DXA) in selected participants
Changes in lipids | 4-month and 1-year
  Total-cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides (mmol/l)
Changes in blood pressure | 4-month and 1-year
  Systolic and diastolic blood pressure (mm/Hg)
Changes in glucose parameters | 4-month and 1-year
  HbA1c (mmol/mol)
Changes in CRP | 4-month and 1-year
  CRP (mg/L)
Changes in Health Related Quality of Life 1 | 4-month and 1-year
  Generic questionnaire: Short Form-36 Health Survey, SF36. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores for each of the 8 domains and summary scores for physical and mental health will be calculated
Changes in Health Related Quality of Life 2 | 4-month and 1-year
  Obesity specific questionnaire: IWQOL-lite. The IWQOL-Lite is a 31-item measure of weight-related quality of life. There are five domain scores (Physical Function, Self-Esteem, Sexual Life, Public Distress and Work) and a total score. Scores for all domains and total score range from 0-100, with lower scores indicating greater impairment.
Changes in Health Related Quality of Life 3 | 4-month and 1-year
  Weight-related Symptom Measure (WRSM). The validated obesity specific WRSM measures 20 symptoms commonly related to being overweight or obese, including foot problems, joint pain, sensitivity to cold, shortness of breath, etc. using two different sets of items. The first set assesses whether or not a patient is experiencing specific symptoms, and the second set rates the level of the distress of the symptoms with values from zero ("not at all") to six ("bothers a very great deal"). The first set creates an additive scale summing symptoms from 0-20, while the second forms a symptom distress scale ranging from 0-120.
Changes in symptoms of depression and anxiety | 4-month and 1-year
  Hospital Anxiety and Depression Scale (HADS). The validated generic HADS measures symptoms of anxiety and depression using 14 items scored from 0-3 It is decomposed into two domains measuring depression (HADS-D) and anxiety (HADS-A), both consisting of seven items yielding a score from 0-21.
Changes in eating behavior | 4-month and 1-year
  The Three Factor Eating Questionnaire -R 21 (TFEQ-R21) measures eating behaviour and has been validated for use in individuals with obesity and will be used in the study. It consists of 21 items comprising three domain scores; (1) uncontrolled eating; assessing the tendency to lose control over eating when feeling hungry or when exposed to external stimuli, (2) cognitive restraint; assessing the conscious restriction of food intake to control body weight or body shape, and (3) emotional eating; assessing overeating related to negative mood states. The domain scores were transformed to 0-100 scales to facilitate comparison; a higher score indicates more uncontrolled, restraint, or emotional eating.
Change in weight from baseline to 4 months | 4-month
  Percent total body weight loss (%TBWL) at 4 months follow-up
Proportions of participants with a TBWL of ≥ 5%, ≥10% and ≥15% at 52-week | 1-year
  TBWL of ≥ 5%, ≥10% and ≥15% at 52-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jøran Hjelmesæth, Professor, Principal Investigator — The Hospital of Vestfold
Locations (1):
- Vestfold Hospital Trust, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No